CLINICAL TRIAL: NCT04272645
Title: A Phase II Multi-Center Trial of Abemaciclib With or Without Atezolizumab in Metastatic Castration Resistant Prostate Cancer
Brief Title: Abemaciclib With or Without Atezolizumab in Metastatic Castration Resistant Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Coordinating site change
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2019.124; HUM00171336 (Other: University of Michigan)
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abemaciclib; atezolizumab; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A - Abemaciclib 200 mg (Experimental): Abemaciclib twice daily. 1 cycle of treatment is 21 days in length.
  Interventions: Drug: Abemaciclib 200 MG
- Arm B - Abemaciclib 150 mg + atezolizumab (Experimental): Atezolizumab on the first day of each 21-day cycle in combination with abemaciclib twice daily.
  Interventions: Drug: Atezolizumab 1200 MG in 20 ML Injection; Drug: Abemaciclib 150 MG
- Experimental: Arm C - Patients with CDK12 loss (Experimental): Group 1 - Atezolizumab: Patients with CDK12 loss will receive atezolizumab monotherapy on the first day of each 21-day cycle
  Group 2 - Abemaciclib 150 mg + atezolizumab: Patients with CDK12 loss will receive atezolizumab on the first day of each 21-day cycle in combination with abemaciclib twice daily.
  Interventions: Drug: Atezolizumab 1200 MG in 20 ML Injection; Drug: Abemaciclib 150 MG

INTERVENTIONS:
Drug: Abemaciclib 200 MG — 200 MG orally BID Days 1-21
  Arms: Arm A - Abemaciclib 200 mg
Drug: Atezolizumab 1200 MG in 20 ML Injection — 1200 mg IV on Day 1 of 21-day cycle
  Arms: Arm B - Abemaciclib 150 mg + atezolizumab; Experimental: Arm C - Patients with CDK12 loss
Drug: Abemaciclib 150 MG — 150 MG orally BID Days 1-21
  Arms: Arm B - Abemaciclib 150 mg + atezolizumab; Experimental: Arm C - Patients with CDK12 loss

SUMMARY:
This research is studying two experimental drugs, abemaciclib and atezolizumab, alone and in combination with each other, to learn about the safety and effectiveness of these treatments and their side effects. This is an investigational study treatment for adult men with metastatic castrate resistant prostate cancer (mCRPC) who have progressive disease despite previous treatment with androgen deprivation therapy (ADT). One group of men (men without a genetic mutation called "CDK12 loss") will receive abemaciclib therapy alone. Two other groups of men (men with CDK12 loss in one group and men without CDK12 loss in the other) will receive the combination of abemaciclib and atezolizumab. Another group of men with CDK12 loss will receive atezolizumab therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic castration resistant prostate cancer (mCRPC), with histologic confirmation of adenocarcinoma of the prostate, without evidence of small cell carcinoma.
* ECOG performance status of 0 or 1.
* Evaluable for response based on: baseline PSA ≥ 2 ng/mL OR measurable disease per RECIST 1.1 criteria.
* Past progression or intolerance to at least one novel antiandrogen therapy (abiraterone, enzalutamide, galeterone, apalutamide, darolutamide, orteronel, seviteronel or equivalent) in either the hormone-sensitive or castration-resistant disease setting.
* Not a candidate for docetaxel or cabazitaxel chemotherapy due to: progression within 12 months of completion or intolerance to prior taxane OR refusal of taxane OR contraindication to, or lack of fitness for taxane OR Investigator assessment that taxane is not clinically indicated or preferred.
* Maintenance of castration status, defined as serum testosterone level of less than 50 ng/dL. Patients must be surgically castrate or maintained on LHRH agonist or antagonist therapy for the duration of the study period.
* Must have recovered from any treatment-related toxicities to ≤ CTCAE grade 1. Patients with ≤ CTCAE grade 2 anorexia, alopecia, neuropathy, and/or fatigue however, are also permitted to enroll.
* Adequate bone marrow, renal, and liver function with no lab abnormalities > CTCAE grade 1. Platelet count of ≥100 x 109 /L.
* Life expectancy of at least 6 months, as determined by a study Investigator.
* Ability to swallow oral medications.
* Ability to understand and willingness to sign an IRB-approved informed consent.

For inclusion specifically in Arm C, documentation (via CLIA approved, CAP certified next generation sequencing [NGS] assay report) of genomic aberration resulting in CDK12 loss of function in metastatic tumor tissue.

Exclusion Criteria:

* Clinical evidence of, or known and untreated metastatic CNS disease.
* Concurrent active malignancy. Patients with non-melanomatous skin cancer, cancer not needing active therapy for at least 2 years, cancer for which the treating investigator deems the subject to be in remission, or any prior malignancy that was treated with curative intent (no evidence of disease for at least 3 years) are also permitted to enroll.
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to planned cycle 1 day 1 of study treatment.
* Patients who have received oral anti-neoplastic intervention such as an oral hormonal agent, PARP inhibitor, AR targeted therapy, or oral experimental agent within 14 days prior to planned cycle 1 day 1 of study treatment.
* Prior treatment with an inhibitor of CDK4 and/or 6.
* Prior treatment with an inhibitor of PD-1, PD-L1, or PD-L2.
* Patients on concurrent therapy with a moderate or strong CYP3A4 inducer or inhibitor which cannot be safely stopped at least five half-lives prior to initiation of therapy with abemaciclib.
* Evidence of an active autoimmune disease that has required systemic treatment within the last 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Patients with conditions requiring replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) are permitted to enroll.
* Live vaccine within 30 days of registration.
* Evidence of active, non-infectious pneumonitis. Patients with a history of asymptomatic radiation pneumonitis with no signs of active process are permitted to enroll.
* Active bacterial or fungal infection, or known detectable viral infection (e.g., Human Immunodeficiency Virus [HIV] or viral hepatitis).
* Arterial or venous thromboembolic event within the last 3 months.
* Significant infection, medical condition, or social situation which, in the opinion of the investigator, would preclude participation or limit the patient's ability to comply with study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) (Arms A and B) | 6 months after start of treatment
  Percentage of patients without disease progression at 6 months after start of treatment. Disease progression as defined by Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria.
Incidence of dose limiting toxicities (DLTs) of combination therapy with abemaciclib and atezolizumab | From start of treatment to end of cycle 1; up to 21 days
  Dose safety for the combination of abemaciclib and atezolizumab is the DLT incidence in Arm B and the combination-therapy cohort of Arm C. DLT is defined in the protocol.

SECONDARY OUTCOMES:
Objective response rate (ORR) (Arms A and B) | Up to 2 years after end of treatment or until study closes, whichever is earliest
  The percentage of patients with at least 50% decline in PSA from pretreatment baseline per PCWG3 criteria
Clinical benefit rate (CBR) (Arms A and B) | Up to 2 years after end of treatment or until study closes, whichever is earliest
  CBR as estimated by proportion of evaluable patients who had complete response (CR), partial response (PR) or stable disease (SD) as their best response to treatment by PCWG3 criteria.
Duration of response (DOR) (Arms A and B) | Up to 2 years after end of treatment or until study closes, whichever is earliest
  DOR among responders by PCWG3 criteria will be reported by treatment arm using Kaplan-Meier methods.
Duration of therapy (DOT) (Arms A and B) | Up to 2 years after end of treatment or until study closes, whichever is earliest
  DOT among responders by PCWG3 criteria will be reported by treatment arm using Kaplan-Meier methods.
Time to progression (TTP) (Arms A and B) | Up to 2 years after end of treatment or until study closes, whichever is earliest
  TTP among responders by PCWG3 criteria will be reported by treatment arm using Kaplan-Meier methods.
Number and severity of Adverse Events of Special Interest (AESI) (all arms) | Up to 2 years after end of treatment or until study closes, whichever is earliest
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) 5.0. Results will be submitted in tabular format, showing the number of each AESI by grade (names of AESI in rows; grades 1 - 5 in columns). AESIs are protocol-specific (as defined in the protocol).
Overall survival among all patients (Arms A and B) | Up to 2 years after end of treatment or until study closes, whichever is earliest
  Number of patients (in arms A and B) alive at 2 years after the end of their treatment.
Overall survival among patients who respond to treatment (Arms A and B) | Up to 2 years after end of treatment or until study closes, whichever is earliest
  Number of patients who responded to treatment (per PCWG3 criteria) alive at 2 years after the end of their treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ajjai Alva, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (4):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University - St. Louis, St Louis, Missouri
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No